CLINICAL TRIAL: NCT03283202
Title: A Phase 1/2 Open-Label Multicenter Study of Avadomide (CC-122) in Combination With R-CHOP-21 for Previously Untreated Poor Risk (IPI>=3) Diffuse Large B-Cell Lymphoma
Brief Title: Study of Safety and Efficacy of Avadomide (CC-122) Combined With RCHOP for Newly-diagnosed DLBCL With Poor Risk Factors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-122-DLBCL-002; U1111-1201-1994 (Registry Identifier: WHO); 2016-003778-42 (EudraCT Number)
Record Dates: First submitted 2017-09-06; First posted 2017-09-14 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Diffuse B-Cell Lymphoma
Keywords: Diffuse B-Cell Lymphoma; R-CHOP-21; International Prognostic Index (IPI)
MeSH Terms: interventions — 3-(5-amino-2-methyl-4-oxoquinazolin-3(4H)-yl)piperidine-2,6-dione; Rituximab; Cyclophosphamide; Vincristine; Prednisone; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Avadomide (CC-122) plus R-CHOP-21 (Experimental): Avadomide (CC-122) by mouth (PO) at varying dose levels (Ph 1) on Days 1 through 5 and Days 8 through 12 plus Rituxan 375 mg/m2 by intravenous (IV) infusion, cyclophosphamide 750mg/m2 by IV infusion, doxorubicin 50 mg/m2 IV, vincristine 1.4 mg/m2 (max is 2.0 mg) IV and 100 mg PO prednisone/prednisolone on Days 1 through 5 of each 21-day treatment cycles for up to 6 total treatment cycles (approximately 18 weeks or 4 months)
  Interventions: Drug: Avadomide (CC-122); Drug: Rituximab; Drug: Cyclophosphamide 750mg/m2 by IV infusion; Drug: Vincristine; Drug: Prednisone

INTERVENTIONS:
Drug: Avadomide (CC-122) — Avadomide (CC-122) by mouth at the assigned dose in Ph 1 starting on Day 1 for 5 consecutive days per week, followed by 2 days without avadomide (CC-122) administration (5/7) for the first two weeks of a 21-day treatment cycle. If the highest proposed dose level to be explored in Phase 1 is applied, the dosing regimen will be 5/7 days for all 3 weeks of each 21-day treatment cycle.
Drug: Rituximab — Rituxan 375 mg/m2 on Day 1 by intravenous (IV) infusion of a 21-day treatment cycle for up to a total of 6 cycles
  Other Names: Rituxan, MabThera
Drug: Cyclophosphamide 750mg/m2 by IV infusion — Cyclophosphamide 750mg/m2 on Day 1 by IV infusion of a 21-day treatment cycle for up to a total of 6 cycles
Drug: Vincristine — Vincristine 1.4 mg/m2 (maximum of 2.0 mg total) on Day 1 by IV bolus on Day 1 of a 21-day treatment cycle for up to a total of 6 cycles
  Other Names: Oncovin, Vincasar
Drug: Prednisone — Prednisone 100 mg PO on Days 1 through 5 of each 21-day treatment or 100mg IV on Day 1 is also acceptable for up to a total of 6 cycles
  Other Names: Prednisolone

SUMMARY:
This is Phase 1/2 study of avadomide (CC-122) in combination with rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone (R-CHOP) chemotherapy, for first-line treatment of patients with Diffuse B-Cell Large B-Cell Lymphoma (DLBCL) that has poor risk factors. Approximately 40% of patients diagnosed with DLBCL are not cured with R-CHOP alone and would need additional treatment for DLBCL in the future. The addition of the experimental drug avadomide (CC-122) with R-CHOP could help in controlling DLBCL in this patient population.

DETAILED DESCRIPTION:
This research study is for patients who have been newly diagnosed with diffuse large B-cell lymphoma DLBCL and are receiving treatment for the first time.

This study will be conducted in two phases. Phase 1 will test the safety of increasing dose levels of avadomide (CC-122) when given in combination with R-CHOP-21 therapy to identify an appropriate dose and schedule for further evaluation in Phase 2. Phase 2 will evaluate the rate of complete response when adding avadomide (CC-122) to the R-CHOP-21 regimen in first-line treatment of patients with poor risk DLBCL.

This study is separated into three periods: the Screening period, the Treatment period and the Follow-up period. Before the patient can receive the drug the doctor will perform test to find out whether he/she can participate in the study. This is done during the Screening period. If the patient and the treating physician determine that the patient is eligible to participate in the study, the patient will be registered in the study and receive avadomide (CC-122) combined with R-CHOP.

In the Treatment period the patient will receive treatment for up to 6 treatment cycles. Each treatment cycle is 21 days long. The full length of the treatment period will be approximately 4 months.

The follow-up period begins when the patient has completed treatment or is discontinued for any reason. During the follow-up period the patient will have fewer exams, test and visits. The first follow-up visit will be 28 days after treatment is completed or discontinued. After that, the follow-up visits will be every 3 months during the first year, then every 6 months until the study is closed.

Upon completion of the Phase 1 portion of the study, a decision not to proceed with the Phase 2 portion was taken by the Sponsor. The decision to terminate the study after Phase 1 was not based on any safety concerns that posed an unacceptable risk for this patient population and no safety issues have been identified

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years of age at the time of signing the informed consent form (ICF).

2. Subject has documented, histologically locally confirmed, previously untreated CD20+ DLBCL (NOS) and the following histologies; refer to the World Health Organization (WHO) 2016 classification (Appendix G):

1. DLBCL associated with chronic inflammation
2. Epstein-Barr virus positive (EBV+) of the elderly
3. T-cell/histiocyte-rich DLBCL 3. Subject is considered an appropriate candidate (per Investigator assessment) for induction therapy with 6 cycles of R-CHOP-21 immunochemotherapy.

   4. Subject has a performance status (PS) of 0-2 according to the Eastern Cooperative Oncology Group (ECOG) scale. Subjects with ECOG PS of 3 may be included if decreased PS is secondary to DLBCL only, and not to comorbidities.

   5. Subject has poor-risk disease defined as International Prognostic Index (IPI) score ≥ 3 (high-intermediate or high-risk classification) and has an age-adjusted IPI defined as ≤ 60 age-adjusted IPI score of 2 with elevated LDH are eligible.

   6. Subject has measurable disease on cross-sectional imaging by computed tomography (CT) with at least one (post-biopsy) measurable lesion ≥ 2.0 cm in its longest dimension.

   7. Subject must appropriately be able to complete Screening assessments before beginning treatment for DLBCL, in the judgement of the Investigator.

   For subjects with bulky disease, B-symptoms, compressive disease, elevated bilirubin due to lymphoma, rapidly progressing adenopathies, or worsening performance status, pre-phase treatment with up to 100 mg/day prednisone, or equivalent, for a maximum of 10 days is permitted prior to beginning the treatment period, at the discretion of the Investigator. A washout period is not required, however, the Screening positron emission tomography (PET), CT, tumor biopsy (if needed), and bone marrow biopsy (if needed) should be completed before initiating corticosteroids.

   8. Subject's central laboratory values must fulfill the following requirements during Screening: Blood product transfusions and hematopoietic growth factors may not be used to meet eligibility criteria. Screening samples should not be collected within 14 days after subject receives a blood product transfusion or growth factors.

   If treatment needs to be urgently started and screening central laboratory results are not available then local laboratory results may be used to confirm eligibility. In these cases, the Celgene medical monitor must be consulted prior to beginning treatment. The investigator must still ensure that samples for the central laboratory are drawn before investigational product is administered and sent to the central laboratory.

   1. Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3 (1.5 x 109/L) unless secondary to extensive bone marrow involvement by lymphoma (ie, ≥ 50%) as demonstrated by unilateral bone marrow core biopsy performed during Screening or within 3 months prior to signing the ICF. In the case of documented extensive bone marrow involvement an ANC ≥ 1,000 cells/mm3 (1.0 x 109/L) is required.

   2. Platelet count ≥ 100,000/mm3 (100 x 109/L) unless secondary to extensive bone marrow involvement by lymphoma (ie, ≥ 50%) as demonstrated by unilateral bone marrow core biopsy performed during Screening or within 3 months prior to signing the ICF. In the case of documented extensive bone marrow involvement, a platelet count of ≥ 75,000/ mm3 (75 x 109/L) is required.

   3. Serum aspartate transaminase (AST/SGOT) or alanine transaminase (ALT/SGPT) ≤ 3.0 x upper limit of normal (ULN). In the case of documented liver involvement by lymphoma, ALT/SGPT and AST/SGOT must be ≤ 5.0 x ULN.

   4. Serum total bilirubin ≤ 2.0 mg/dL (34 μmol/L). In the case of Gilbert's syndrome, or documented liver or pancreatic involvement by lymphoma, serum total bilirubin must be ≤ 5.0 mg/dL (86 μmol/L).

   5. Calculated creatinine clearance (CrCl) of ≥ 50 mL/min by the Cockcroft-Gault formula.

   9. Subject must understand and voluntarily sign an Informed Consent Form (ICF) prior to any study-specific assessments/procedures being conducted.

   10. Subject is willing and able to adhere to the study visit schedule and other protocol requirements.

   11. Sufficient tissue from diagnostic tumor/ lymph node biopsy (from within 2 months prior to ICF signature) must be available for translational research purposes or subject is willing to undergo core needle or incisional/ excisional biopsy during Screening.

   12. Females of childbearing potential (FCBP)1 must:
   1. Agree to use two reliable forms of contraception simultaneously or to practice complete abstinence (True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence [eg calendar, ovulation, symptothermal or post-ovulation methods] and withdrawal are not acceptable methods of contraception.) from heterosexual contact during the following time periods related to this study: 1) for at least 28 days before starting avadomide (CC-122); 2) while taking avadomide (CC-122); 3) during dose interruptions; and 4) for at least 28 days after the last dose of avadomide (CC-122) as specified in the Pregnancy Prevention and Risk Management Plan (PPRMP)
   2. Have a negative result confirmed for a medically supervised urine (or serum) pregnancy test (with a sensitivity of at least 25 mIU/mL) 10-14 days prior to the first dose of IP. A second pregnancy test performed within 24 hours prior to the first dose of IP must also be confirmed to be negative prior to IP administration.

      * If urgent treatment is needed and requires a shorter window of screening, please immediately contact the medical monitor

   13. Avoid conceiving for at least 12 months after the last dose of rituximab, or according to the local rituximab Prescribing Information or Summary of Product characteristics (SmPC); at least 28 days after the last dose of any other study drug.

   1. Agree to ongoing pregnancy testing during the course of the study as outlined in the PPRMP.

   14. Male subjects must:
   1. Practice complete abstinence (True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence [eg calendar, ovulation, symptothermal or post-ovulation methods] and withdrawal are not acceptable methods of contraception.) or agree to use a condom during sexual contact with a pregnant female or a FCBP for at least 12 months after the last dose of rituximab.
   2. Agree to not donate semen or sperm for at least 12 months following the last dose of rituximab.

   15. All subjects must:
   1. Understand that avadomide (CC-122) could have a potential teratogenic risk.
   2. Agree to abstain from donating blood while taking IP and for at least 28 days following discontinuation of IP.
   3. Agree not to share IP with another person
   4. Be counseled about pregnancy precautions and risks of fetal exposure and agree to requirements of the Pregnancy Prevention and Risk Management Plan (PPRMP)

   16. Subject is able to swallow pills.

   Exclusion Criteria:

   1. Subject is seropositive for or has active viral infection with hepatitis B virus (HBV):
   1. HBV surface antigen (HBsAg) positive
   2. HBV surface antigen (HBsAg) negative, HBV surface ant ibody (ant i-HBs) posit ive and/or HBV core antibody (ant i-HBc) positive, and detectable viral DNA Subjects who are seropositive because of prior HBV vaccination are eligible (anti- HBs positive, anti-HBc negative, and HBsAg negative).

   2. Subject is known to be seropositive for, or have an active infection with, hepatitis C virus (HCV).

   3. Subject is known to be seropositive for, or have an active infection with, human immunodeficiency virus (HIV).

   4. Subject has any neuropathy > Grade 1. 5. Subject has impaired cardiac function or clinically significant cardiac diseases, including any of the following:
   1. Left ventricular ejection fraction (LVEF) < 45% as determined by multi-gated acquisition scan (MUGA) or echocardiogram (ECHO).
   2. Complete left bundle branch or bifascicular block.
   3. Persistent or clinically meaningful ventricular arrhythmias.
   4. Unstable angina pectoris or myocardial infarction ≤ 3 months prior to starting treatment in the study.
   5. Troponin-T value > 0.4 ng/mL or B-type natriuretic protein (BNP) > 300 pg/mL by central laboratory assessment Subjects with baseline troponin-T > ULN or BNP > 100 pg/mL are eligible but must have a cardiologist evaluation prior to enrollment in the trial for baseline assessment and optimization of cardioprotective therapy.

      If troponin-T is not usually tested by local laboratory then troponin-I may be used to confirm subject meets the Screening eligibility criteria. The central laboratory sample must still be collected prior to first dose and sent to central laboratory. Elevated cut-off value for troponin I will depend on the assay used at the site. If baseline troponin I >ULN, the subject must have a cardiologist consultation prior to enrollment and optimization of cardioprotective therapy.

      In case of discrepancy between both troponin-I and troponin-T test, the troponin-T test will be repeated.
   6. Subject has confirmed central nervous system (CNS) involvement by DLBCL. Subjects at risk for CNS involvement per Investigator assessment must receive prophylaxis. For subjects at risk, or with any neurological symptoms, testing for CNS involvement is required at Screening.
   7. Subject has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
   8. Subject has any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
   9. Subject has any condition that confounds the ability to interpret data from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2020-12-16 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose/Maximum Administered Dose (MTD/MAD) (Phase 1) | Through 6 cycles of treatment (approximately 18 weeks or 4 months)
  Frequency of dose-limiting toxicities (DLTs) associated with the addition of avadomide (CC-122) to R-CHOP-21 therapy
Complete Response Rate (CRR); Percentage of participants experiencing positron emission tomography (PET)-negative complete response (CR) (Phase 2) | 6 to 8 weeks after completion of treatment
  CR is defined as target nodes/nodal masses regress to ≤ 1.5 cm in LDi; no extralymphatic sites of disease; no measurable lesions, no organ enlargement and normal morphology on bone marrow (BM) exam; immunohistochemically (IHC) negative

SECONDARY OUTCOMES:
Overall Response Rate (ORR); Percentage of participants who achieve a PR or CR according to the Lugano criteria. | 6 to 8 weeks after completion of treatment
  ORR is defined as the rate of the responses (including CR; see definition above for CR and PR; PR is defined as ≥ 50% decrease in sum of perpendicular diameters (SPD) of up to 6 target measurable nodes and extranodal sites. When a lesion is too small to measure on CT, assign 5 mm × 5 mm as the default value; When no longer visible, 0 × 0 mm; for a node > 5 mm × 5 mm, but smaller than normal, use actual measurement for calculation; Absent/normal, regressed, but no increase in non measurable lesions; spleen must have regressed > 50% in length beyond normal and no new lesions.
ORR by Predictive Gene Signature | 6 to 8 weeks after completion of treatment
  ORR by Predictive Gene Signature is defined as the correlation between baseline gene expression signatures and clinical response to study treatment
Progression-free Survival (PFS) | From enrollment up to 24 months after last subject is enrolled
  PFS is defined as the time from enrollment to disease progression or death from any cause
Event-free Survival (EFS) | At 12 and 24 months after enrollment
  EFS is defined as the percentage of participants without event (relapse or progression, unplanned re-treatment of lymphoma after initial immunochemotherapy, or death from any cause)
Overall Survival (OS) | Up to 24 months after enrollment
  OS is defined as the time from enrollment until death from any cause
Adverse Events (AEs) | From enrollment until at least 28 days after completion of study treatment
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, including laboratory test values, regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a pre- existing condition) should be considered an AE.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Delarue, MD, Study Director — Celgene
Locations (15):
- United States (3):
  - George Washington University, Washington D.C., District of Columbia
  - Moffitt Cancer Center, Tampa, Florida
  - Washington University, St Louis, Missouri
- Belgium (2):
  - UZ Gent, Ghent
  - University Hospital Gasthuisberg, Lueven
- Canada (3):
  - Tom Baker Cancer Center, Calgary, Alberta
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- Spain (7):
  - Hospital Germans Trias I Pujol, Badalona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital de San Pedro de Alcantara, Cáceres
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen Del Rocio, Seville

IPD SHARING:
Plan to Share IPD: Undecided